CLINICAL TRIAL: NCT00141167
Title: A Twelve-Week, Double-Blind, Placebo-Controlled, Multicenter Study With Follow-up Evaluating the Safety and Efficacy of Varenicline Tartrate 1 MG BID for Smoking Cessation
Brief Title: A Twelve-Week Study of Varenicline for Safety and Efficacy in Comparison With Placebo for Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051045; NCT00155298 (obsolete NCT alias)
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

INTERVENTIONS:
Drug: varenicline

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of varenicline given for a twelve week treatment period in comparison with placebo for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have smoked an average of at least 10 cigarettes per day during the past year and over the month prior to the screening visit, with no period of abstinence greater than 3 months in the past year.

Exclusion Criteria:

* Subjects who have used bupropion, Zyban, or Wellbutrin previously.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2005-02; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
4 week continuous quit rate ( 4 week CQR ) for weeks 9 -12

SECONDARY OUTCOMES:
Continuous abstinence rate weeks 9-24
Long-term Quit Rate at week 24
7 day point prevalence week 12 and 24
Results of Minnesota Nicotine Withdrawal Scale
Brief Questionnaire of Smoking Urges
Smoking Effects Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- South Korea (3):
  - Pfizer Investigational Site, Anyang-si, Gyeonggi-do
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Seoul
- Taiwan (5):
  - Pfizer Investigational Site, Kweishan, Taoyuan County
  - Pfizer Investigational Site, Hualien City
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Tsai ST, Cho HJ, Cheng HS, Kim CH, Hsueh KC, Billing CB Jr, Williams KE. A randomized, placebo-controlled trial of varenicline, a selective alpha4beta2 nicotinic acetylcholine receptor partial agonist, as a new therapy for smoking cessation in Asian smokers. Clin Ther. 2007 Jun;29(6):1027-39. doi: 10.1016/j.clinthera.2007.06.011. PMID 17692719